CLINICAL TRIAL: NCT05268159
Title: Neural Basis of Unilateral Spatial Neglect After Stroke: a Retrospective Disconnectome Based Study
Brief Title: Disconnection and Unilateral Spatial Neglect
Acronym: DISCONEGLECT
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: HLJ_2022_02
Record Dates: First submitted 2022-02-24; First posted 2022-03-07 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-02

CONDITIONS: Stroke
Keywords: Stroke; Unilateral spatial neglect; MRI; Disconnectome,; Cognition
MeSH Terms: conditions — Stroke | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stroke patients: Stroke patients admitted to the Lille Neurological rehabilitation unit after a first-ever hemispheric stroke, assessed at the subacute phase (< 6months)
  Interventions: Other: Cognitive assessment

INTERVENTIONS:
Other: Cognitive assessment — Assessment of unilateral spatial neglect, attention, executive functions and memory

SUMMARY:
Retrospective cohort study of consecutive patients investigated in a neurorehabilitation ward after a first hemispheric stroke. Unilateral spatial Neglect (USN) and other cognitive impairments (including attention, executive functions, memory) have been assessed in routine care at the subacute phase (<6 months). MRI scans have also been done in routine care.

The study aims at linking lesion characteristics, disconnections induced and expression of the different modalities of USN

ELIGIBILITY:
Inclusion Criteria:

* First hemispheric adult stroke patient
* Non-opposed to inclusion
* Confirmed by MRI
* Assessment of cognitive functions during the subacute phase (3 weeks to 6 months after stroke onset

Exclusion Criteria:

* History of previous stroke or neurological disorders
* Inability to perform cognitive assessment due to severe comprehension, cognitive or psychiatric disorder
* Uncorrected severe loss of visual acuity
* Contra-indications to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients admitted in neurorehabilitation ward after first hemispheric stroke
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2011-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Assessment of peripersonal Unilateral Neglect with the BEN (Batterie d'évaluation de la negligence, Battery of tests for the quantitative assessment of unilateral neglect) | One assessment, during the subacute phase after stroke (3 weeks to 6 months)

SECONDARY OUTCOMES:
Assessment of personal Unilateral Spatial Neglect with the Fluff Test | One assessment, during the subacute phase after stroke (3 weeks to 6 months)
Assessment of personal Unilateral Spatial Neglect with the Comb and Razor Test | One assessment, during the subacute phase after stroke (3 weeks to 6 months)
Assessment of Attention with the Test of Attentional Performance | One assessment, during the subacute phase after stroke (3 weeks to 6 months)
Assessment of Executive Functions with the Stroop Test | One assessment, during the subacute phase after stroke (3 weeks to 6 months)
Assessment of Executive Functions with the Trail Making Test | One assessment, during the subacute phase after stroke (3 weeks to 6 months)
Assessment of Executive Function with Verbal and Categorial Fluency test | One assessment, during the subacute phase after stroke (3 weeks to 6 months)
Assessment of Executive Functions with the test of commissions | One assessment, during the subacute phase after stroke (3 weeks to 6 months)
Assessment of verbal Memory with the verbal span task | One assessment, during the subacute phase after stroke (3 weeks to 6 months)
Assessment of verbal Memory with the Grober and Buschke Task | One assessment, during the subacute phase after stroke (3 weeks to 6 months)
Assessment of visual Memory with the Doors test | One assessment, during the subacute phase after stroke (3 weeks to 6 months)
Assessment of visual Memory with the Rey figure test | One assessment, during the subacute phase after stroke (3 weeks to 6 months)
Identification of brain lesions by Anatomical MRI (T1, FLAIR, T2*, Diffusion) | up to 6 months
Postural assessment with the PASS | 1 month after stroke
Postural assessment with the PASS | 3 months after stroke
Gait assessment (Lindmark score) | 1 month after stroke
Gait assessment (Lindmark score) | 3 months after stroke

CONTACTS AND LOCATIONS:
Overall Officials: Etienne Allart, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Swynghedauw, Lille, France